CLINICAL TRIAL: NCT06596629
Title: Nerve Transfers (reinnervation of the Posterior Interosseus Nerve and Anterior Interosseus Nerve) in Patients with Cervical Spinal Cord Injury: Duration Until Effect, Influence of Age and Impact of Time to Surgery on the Effect
Brief Title: Nerve Transfers for Restoration of Hand Function in Cervical Spinal Cord Injury: Effects and Influencing Factors
Status: Completed | Type: Observational
Sponsor: Roessingh Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-17418
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Nerve Transfer
Keywords: spinal cord injury; tetraplegia; posterior interosseus nerve; anterior interosseus nerve; hand function
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about influencing factors on the clinical outcomes of nerve transfers used to restore hand function in patients with cervical spinal cord injury (CSCI). Specifically, the study focuses on the reinnervation of the posterior interosseus nerve (PIN) and the anterior interosseus nerve (AIN).

The main questions it aims to answer are:

1. What is the duration after nerve transfer surgery until effect is achieved?
2. What is the influence of the participants age during surgery on the effect of a nerve transfer?
3. What is the impact of time interval from the date of spinal cord injury to the date of nerve transfer surgery?

Participants are not directly involved in this study since data will be retrospectively collected from the Electronic Patients Records (EPD).

DETAILED DESCRIPTION:
Spinal cord injury (SCI) has a profound impact on the quality of life. Patients with a cervical spinal cord injury (CSCI) additionally suffer from upper extremity impairments, leading to increased dependence on others for daily life activities and a further decline in quality of life. For many patients, improvement of hand function is therefore the highest-ranked goal in rehabilitation after CSCI. Conventionally, tendon transfers have been widely used to reconstruct upper extremity function. Over the past decade, there has been growing interest in employing nerve transfer techniques for reconstruction of upper limb function in tetraplegia. Specifically for reconstruction of hand function, reinnervation of the posterior interosseus nerve (PIN) provides restoration of extension of fingers and thumb, while reinnervation of the anterior interosseus nerve (AIN) is intended to restore flexion of thumb, index finger and middle finger.

Since previous studies already reported success rates for the different nerve transfers, this study will mainly focus on the factors influencing the clinical outcomes of the reinnervation of PIN and AIN in patients with cervical spinal cord injury. Specifically, the study will focus on the impact of age during surgery and the interval between spinal cord injury and surgery on clinical outcomes.

In this single-center retrospective case series, data will be collected from patients with a cervical spinal cord injury who underwent single or multiple nerve transfers in one or both upper limbs to reanimate the PIN and/or AIN. Informed consent is not required, as this study involves a retrospective analysis of anonymized data without any direct intervention or interaction with patients.

Data will be extracted from the Electronic Patient Records (EPD) at Roessingh. This data will be anonymized, by using exclusive numbers for all patients. The identifying information will be kept in a separate list only accessible by the lead researcher. In all analyses, only the patient specific codes will be used.

Baseline data will include age, gender and smoking habits. SCI related data compromises the date of injury, mechanism of injury, neurological level, motor level, grade of International Classification of Surgery of the Hand in Tetraplegia (ICSHT) and the American Spinal Injury Association (ASIA) grade. The specific surgeries performed and their dates will be recorded. Patients records will be reviewed to determine the dates of when the effect of nerve transfers were observed. Additionally, the number of treated limbs and the number of patients with limiting spasticity or restricted range of motion in the hands will be documented.

As this is a retrospective study, some data may be missing, and variables will be reported as such. Data that is uninterpretable will also be reported as missing.

All adverse events and serious adverse events will be recorded.

Statistical analysis: kaplan-Meier survival analysis will be used to estimate the time until effect of nerve transfers occured. Spearman rank correlations will be used to assess the relationship between the variables, specifically between the results of nerve transfers and 'age during surgery' and 'time between spinal cord injury and nerve transfer surgery'.

ELIGIBILITY:
Inclusion Criteria:

* patients with cervical spinal cord injury
* single or multiple nerve transfers in one or both upper limbs to reanimate the posterior interosseus nerve (PIN) or anterior interosseus nerve (AIN).
* Surgery performed in Medical Spectrum Twente (MST) in Enschede.
* Postoperative treatment in Roessingh, Centre for Rehabilitation (RCR) in Enschede.
* Surgeries performed between February 2019 and February 2024.

Exclusion Criteria:

* patients with pre-existing neurological comorbidities

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a cervical spinal cord injury, ≥ 12 years and older, who underwent single or multiple nerve transfers in one or both upper limbs to reanimate the posterior interosseus nerve (PIN) and/or anterior interosseus nerve (AIN).
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Duration until result of nerve transfers | up to 4 weeks
  Defined as the time until 'first result' or 'desired result' is achieved following nerve transfer surgery.
  First result: defined as the first visible muscle contraction in the reinnervated muscles. For the posterior interosseus nerve (PIN), this includes any contraction of thumb and/or finger extension. For the anterior interosseus nerve (AIN), this refers to any visible flexion of thumb, index finger and middle fingers .
  Desired result: for reanimation of the posterior interosseus nerve (PIN), this is defined as the patient's ability to extent the thumb and fingers sufficiently to achieve a desirable hand opening. Successful reinnervation of the anterior interosseus nerve (AIN) will be documented when patients are able to flex the thumb and fingers to form a fist.
  Dates of first result, desired result and date of surgery will be extracted from patient's records.
  Duration after surgery until 'first result' and 'desired result' will be expressed in months.

SECONDARY OUTCOMES:
Age during surgery | Up to 4 weeks
  The influence of age during surgery on the results of nerve transfers will be assessed.
  Patients records will be reviewed to extract the following information: birth date, surgery date and dates of first result en desired result. To determine the age of the patient at the time of surgery, the difference between the date of birth and the date of surgery will be calculated .
  Age during surgery will be expressed in years.
  Hypothesis: younger patients are expected to achieve earlier and better outcomes from nerve transfer surgery.
Time between spinal cord injury and nerve transfer surgery | Up to 4 weeks
  The influence of time to surgery on the results of nerve transfers will be assessed.
  Patient's records will be reviewed to extract the following information: spinal cord injury date, surgery date and dates of first result and desired result. Time between spinal cord injury date and surgery date will be expressed in months.
  Hypotheses: surgeries performed within 12 months after spinal cord injury will result in earlier and better outcomes from nerve transfer surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nora W Jacobs, MD, Study Chair — Roessingh,Centre for Rehabilitation
Locations (1):
- Roessingh, Centre for Rehabilitation, Enschede, Overijssel, Netherlands